CLINICAL TRIAL: NCT00430677
Title: A Phase II/III Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Abatacept Versus Placebo on a Background of Mycophenolate Mofetil and Glucocorticosteroids in Subjects With Active Proliferative Glomerulonephritis Due to Systemic Lupus Erythematosus (SLE)
Brief Title: Efficacy and Safety Study of Abatacept to Treat Lupus Nephritis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated due to failure to meet the primary efficacy endpoint in the Short-term Period
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-075
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Results first posted 2012-05-11 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Adrenal Cortex Hormones; Prednisone; Prednisolone; Abatacept; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Abatacept 30 mg/kg+Corticosteroids+MMF (Experimental): Short-term Period
  Interventions: Drug: Corticosteroids (prednisone or prednisolone); Drug: Abatacept; Drug: Mycophenolate mofetil (MMF)
- Abatacept 10 mg/kg+Corticosteroids+MMF (Experimental): Short-term Period
  Interventions: Drug: Corticosteroids (prednisone or prednisolone); Drug: Abatacept; Drug: Mycophenolate mofetil (MMF)
- Placebo+Corticosteroids+MMF (Experimental): Short-term Period
  Interventions: Drug: Corticosteroids (prednisone or prednisolone); Drug: Mycophenolate mofetil (MMF)
- Abatacept 10mg/kg (Experimental): Long-term Extension Period
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Corticosteroids (prednisone or prednisolone) — tablets, oral, 0.5-0.8 mg/kg, daily
  Arms: Abatacept 10 mg/kg+Corticosteroids+MMF; Abatacept 30 mg/kg+Corticosteroids+MMF; Placebo+Corticosteroids+MMF
Drug: Abatacept — intravenous solution, injectable, 30 mg/kg, every 28 days
  Other Names: Orencia; BMS-188667
  Arms: Abatacept 30 mg/kg+Corticosteroids+MMF
Drug: Abatacept — intravenous solution, injectable, 10 mg/kg, every 28 days
  Other Names: Orencia; BMS-188667
  Arms: Abatacept 10 mg/kg+Corticosteroids+MMF
Drug: Mycophenolate mofetil (MMF) — tablets, oral, 1.5 to 2 g, daily
  Arms: Abatacept 10 mg/kg+Corticosteroids+MMF; Abatacept 30 mg/kg+Corticosteroids+MMF; Placebo+Corticosteroids+MMF
Drug: Abatacept — intravenous solution, injectable, 10 mg/kg, every 28 days
  Arms: Abatacept 10mg/kg

SUMMARY:
The purpose of this clinical research study is to learn if addition of abatacept is safe and improves the effectiveness of treatment of patients with active lupus nephritis who are also taking mycophenolate mofetil (MMF) and corticosteroids.

DETAILED DESCRIPTION:
Double Blind Period: Treatment, Parallel Assignment, Double Blind (Subject, Investigator), Randomized, Active Control, Safety/Efficacy Study

Open Label Period: Prevention, Single Group Assignment, Open Label, Uncontrolled, Safety/Efficacy Study

ELIGIBILITY:
Inclusion Criteria:

* Systemic Lupus Erythematosus (SLE) as defined by meeting at least 4 of the 11 classification criteria of the American College of Rheumatology for the classification of Systemic Lupus Erythematosus, either sequentially or coincident. The 4 criteria need not be present at study entry
* Renal biopsy within 12 months prior to screening visit indicating active proliferative lupus glomerulonephritis (met ISN/RPS Class III or IV classification criteria [2003], excluding Class III [C], IV-S [C] and IV-G [C], or the World Health Organization Class III or IV classification criteria [1982], excluding Class IIIc, IVd). If the renal biopsy was performed >3 months but ≤12 months prior to screening visit, at least 1 of the following 3 serologies (performed locally) must have been abnormal prior to screening visit: complement (C3 or C4) level below normal range OR anti-dsDNA >upper limit of normal range.
* A stable serum creatinine ≤3 mg/dL

Exclusion Criteria:

* Subjects with a rise in serum creatinine of ≥1 mg/dL within 1 month prior to the screening visit
* Subjects with drug-induced SLE, as opposed to idiopathic SLE
* Subjects with severe, unstable and/or progressive Central nervous system (CNS) lupus
* Subjects with autoimmune disease other than SLE as their main diagnosis (e.g.; Rheumatoid arthritis (RA), Multiple Sclerosis [MS])
* Subjects who have received treatment with cyclophosphamide within 3 months of randomization (Day 1).
* Subjects who have received treatment with rituximab < 6 months prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2007-06; Primary Completion 2010-09 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (76):
- United States (14):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Arizona Arthritis Center, Tucson, Arizona
  - Wallace Rheumatic Study Center, Los Angeles, California
  - University Of Kansas Medical Center, Kansas City, Kansas
  - Boston University School Of Medicine, Boston, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Suny Downstate Medical Center, Brooklyn, New York
  - Northshore Lij Health System, Lake Success, New York
  - The Feinstein Institute For Medical Research, Manhasset, New York
  - Suny Upstate Medical University, Syracuse, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Ok Medical Research Foundation, Oklahoma City, Oklahoma
  - Rheumatology Consultants Pllc, Knoxville, Tennessee
  - Virginia Mason Medical Center, Seattle, Washington
- Argentina (4):
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
- Australia (4):
  - Local Institution, Liverpool, New South Wales
  - Local Institution, Clayton, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Parkville, Victoria
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Leuven
- Brazil (5):
  - Local Institution, Goiânia, Goiás
  - Local Institution, Curitiba, Paraná
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, São Paulo, São Paulo
- Canada (4):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Toronto, Ontario
  - Local Institution, Québec, Quebec
- China (4):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Xi’an, Shanxi
- France (4):
  - Local Institution, Créteil
  - Local Institution, Paris
  - Local Institution, Strasbourg
  - Local Institution, Toulouse
- Local Institution, Hong Kong, Hong Kong
- India (9):
  - Local Institution, Gujarat, Ahmedabad
  - Local Institution, Secunderabad, Andhra Pradesh
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Nadiād, Gujarat
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Kochi, Kerala
  - Local Institution, Mumbai, Maharajhsra
  - Local Institution, Hyderabad
  - Local Institution, Visakhapatnam
- Mexico (7):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, San Luis Potosí City, San Luis Potosí
  - Local Institution, Metepec, State of Mexico
  - Local Institution, Mérida, Yucatán
- Poland (3):
  - Local Institution, Bydgoszcz
  - Local Institution, Gdansk
  - Local Institution, Wroclaw
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Yaroslaval
  - Local Institution, Yekaterinburg
- South Africa (3):
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Observatory, Western Cape
  - Local Institution, Panorama, Western Cape
- South Korea (2):
  - Local Institution, Seoul, Sungdong-Gu
  - Local Institution, Seoul
- Taiwan (4):
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Taipei
  - Local Institution, Taoyuan District
- Local Institution, Gaziantep, Turkey (Türkiye)
- United Kingdom (2):
  - Local Institution, Cambridge, Cambridgeshire
  - Local Institution, London, Greater London

REFERENCES:
- [Derived] Wolf BJ, Spainhour JC, Arthur JM, Janech MG, Petri M, Oates JC. Development of Biomarker Models to Predict Outcomes in Lupus Nephritis. Arthritis Rheumatol. 2016 Aug;68(8):1955-63. doi: 10.1002/art.39623. PMID 26867033
- [Derived] Furie R, Nicholls K, Cheng TT, Houssiau F, Burgos-Vargas R, Chen SL, Hillson JL, Meadows-Shropshire S, Kinaszczuk M, Merrill JT. Efficacy and safety of abatacept in lupus nephritis: a twelve-month, randomized, double-blind study. Arthritis Rheumatol. 2014 Feb;66(2):379-89. doi: 10.1002/art.38260. PMID 24504810
- [Derived] Wofsy D, Hillson JL, Diamond B. Comparison of alternative primary outcome measures for use in lupus nephritis clinical trials. Arthritis Rheum. 2013 Jun;65(6):1586-91. doi: 10.1002/art.37940. PMID 23529285
- [Derived] Wofsy D, Hillson JL, Diamond B. Abatacept for lupus nephritis: alternative definitions of complete response support conflicting conclusions. Arthritis Rheum. 2012 Nov;64(11):3660-5. doi: 10.1002/art.34624. PMID 22806274
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 423 participants were enrolled and screened; 300 were randomized. Of the 228 participants who completed the short-term period, 211 received treatment in the long-term extension period. A total of 166 participants (78.7%) remained in the study at the time of study termination by the sponsor.
Groups:
- Abatacept 30/10 mg/kg: Short-term period: Abatacept 30/10 mg/kg regimen by intravenous (IV) infusion: abatacept 30 mg/kg (by weight) on Days 1, 15, 29, and 57, followed by abatacept (fixed dose) approximating 10 mg/kg on Days 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral Mycophenolate mofetil (MMF) and oral prednisone or prednisone-equivalent Long-term extension period: Participants received abatacept in a weight-tiered dose of approximately 10 mg/kg administered every 28 days by intravenous (IV) infusion in addition to oral mycophenolate mofetil (MMF) and oral prednisone or prednisone-equivalent.
- Abatacept 10/10 mg/kg: Short-term period: Abatacept 10/10 mg/kg regimen by IV infusion: abatacept (fixed dose) approximating 10 mg/kg on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent Long-term extension period: Participants received abatacept in a weight-tiered dose of approximately 10 mg/kg administered every 28 days by intravenous (IV) infusion in addition to oral mycophenolate mofetil (MMF) and oral prednisone or prednisone-equivalent.
- Placebo: Short-term period: Placebo (Dextrose 5% in water [D5W]) or Normal Saline (NS) by IV infusion on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent Long-term extension period: Participants received abatacept in a weight-tiered dose of approximately 10 mg/kg administered every 28 days by intravenous (IV) infusion in addition to oral mycophenolate mofetil (MMF) and oral prednisone or prednisone-equivalent.
Period: Short-term Period
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Started | 99 (1 participant died before receiving the first dose of study medication) | 99 (1 participant took infliximab on day 1 and was discontinued before receiving study medication.) | 100
Completed | 76 (Completed the short-term period) | 74 (Completed the short-term period) | 78 (Completed the short-term period)
Not Completed | 23 | 25 | 22
Not completed — Death | 1 | 1 | 5
Not completed — Adverse Event | 15 | 13 | 9
Not completed — Lack of Efficacy | 5 | 6 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Participant no longer met study criteria | 1 | 1 | 2
Not completed — Poor compliance/ noncompliance | 0 | 1 | 0
Not completed — Pregnancy | 0 | 2 | 0
Period: Long-term Extension Period
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Started | 70 | 67 | 74
Completed | 10 (Completed the long-term extension period) | 9 (Completed the long-term extension period) | 11 (Completed the long-term extension period)
Not Completed | 60 | 58 | 63
Not completed — Death | 1 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 5
Not completed — Lack of Efficacy | 5 | 3 | 8
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 1 | 2
Not completed — Pregnancy | 1 | 1 | 0
Not completed — Administrative reason by sponsor | 41 | 49 | 46
Not completed — Other | 2 | 1 | 1
Not completed — Poor compliance/noncompliance | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Abatacept 30/10 mg/kg: Abatacept 30/10 mg/kg regimen by IV infusion: abatacept 30 mg/kg (by weight) on Days 1, 15, 29, and 57, followed by abatacept approximating 10 mg/kg on Days 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent
- Abatacept 10/10 mg/kg: Abatacept 10/10 mg/kg regimen by IV infusion: abatacept approximating 10 mg/kg on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent
- Placebo: Placebo (Dextrose 5% in water [D5W]) or Normal Saline (NS) by IV infusion on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent
- Total: Total of all reporting groups
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo | Total
Number analyzed (Participants) | 99 | 99 | 100 | 298
Age, Customized [Number; unit: Participants]
  16 - 29 years | 55 | 52 | 46 | 153
  30 - 39 years | 28 | 30 | 33 | 91
  40 - 49 years | 10 | 10 | 18 | 38
  50 - 59 years | 5 | 6 | 2 | 13
  >= 60 years | 1 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 86 | 81 | 251
  Male | 15 | 13 | 19 | 47
Race [Number; unit: Participants]
  White | 28 | 45 | 38 | 111
  Black/African American | 6 | 3 | 5 | 14
  American Indian/Alaska Native | 0 | 1 | 0 | 1
  Native Hawaiian/Other Pacific Islander | 1 | 0 | 0 | 1
  Other Asian | 60 | 49 | 55 | 164
  Other | 4 | 1 | 2 | 7
Weight, Group [Number; unit: participants]
  <60 kg | 54 (0.68) | 55 (0.62) | 45 (0.73) | 154
  60 - 100 kg | 42 | 43 | 51 | 136
  >100 kg | 3 | 1 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Time to First Confirmed Complete Renal Response (CRR) During the Short-term (Double-blind) Period
Description: Confirmed at 2 consecutive visits. CRR defined as meeting all of 5 criteria. Renal function (RF): (Glomerular filtration rate [GFR] calculated using Modification of Diet in Renal Diseases equation equation) Calculated function abnormal at screening visit - return of renal function to greater than or equal to 90% of function at approximately 6 months prior to onset of the current episode of lupus nephritis. Calculated function normal at screening visit - estimated renal function 90% or greater of level at screening visit. Proteinuria: urinary protein/creatinine ratio <30 mg/mmol. Hematuria: red blood cell (RBC) count within normal limits of Central Laboratory. Pyuria: White blood cell count (WBC) within normal limits of Central Laboratory. Cylindruria: No RBC or WBC casts reported.
Time Frame: Day 1 (randomization) to 12 months.
Population: All randomized participants who received treatment. Includes participants who died and who were censored at the time of discontinuation.
Measure: Number; unit: days
Groups:
- Abatacept 30/10 mg/kg: Abatacept 30/10 mg/kg regimen by intravenous (IV) infusion: abatacept 30 mg/kg (by weight) on Days 1, 15, 29, and 57, followed by abatacept (fixed dose) approximating 10 mg/kg on Days 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral mycophenolate mofetil (MMF) and oral prednisone or prednisone-equivalent
- Abatacept 10/10 mg/kg: Abatacept 10/10 mg/kg regimen by IV infusion: abatacept (fixed dose) approximating 10 mg/kg on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
days | NA [NE to NE] — The Kaplan-Meier median time to confirmed CRR was not reached due to a small number of events (such as, fewer than 50% of participants achieved confirmed CRR). | NA [NE to NE] — The Kaplan-Meier median time to confirmed CRR was not reached due to a small number of events (such as, fewer than 50% of participants achieved confirmed CRR). | NA [NE to NE] — The Kaplan-Meier median time to confirmed CRR was not reached due to a small number of events (such as, fewer than 50% of participants achieved confirmed CRR).
Statistical Analysis 1: Comparison: Abatacept 30/10 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.746, Regression, Cox — The median time to confirmed CRR was not estimable due to the low number of events. However, the time to confirmed CRR was compared between the abatacept and placebo treatment regimens using a score test; Cox Proportional Hazard = 1.1, 95% CI 2-sided [0.60 to 2.03] — Point estimate, 95% CI and P-value (based on Score Test) for the hazard ratio is determined by a Cox proportional hazards model including treatment as a covariate and stratified by prior treatment status
Statistical Analysis 2: Comparison: Abatacept 10/10 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.118, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Cox Proportional Hazard = 1.6, 95% CI 2-sided [0.89 to 2.83] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With Confirmed Complete Renal Response (CRR) During Short-term Period
Description: as for outcome 1
Time Frame: Day 1 to 12 months
Population: All randomized participants who received treatment. Participants who discontinued early without meeting the confirmed CRR criteria were imputed as nonresponders.
Measure: Number; unit: Participants
Groups:
- Abatacept 30/10 mg/kg: Abatacept 30/10 mg/kg regimen by intravenous (IV) infusion: abatacept 30 mg/kg on Days 1, 15, 29, and 57, followed by abatacept approximating 10 mg/kg on Days 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent
- Abatacept 10/10 mg/kg: Abatacept 10/10 mg/kg regimen by IV infusion: abatacept approximating 10 mg/kg on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral mycofenolate mofetil (MMF) and oral prednisone or prednisone-equivalent
- Placebo: Placebo (dextrose 5% in water) or normal saline by IV infusion on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Participants | 22 | 27 | 20

3. Secondary Outcome: Participants Achieving a Confirmed Complete Renal Response (CRR) at Month 12 During Short-term Period
Description: as for outcome 1
Time Frame: At Month 12 from Day 1
Population: All randomized participants who received treatment. Missing response values were imputed as nonresponders for participants who discontinued early after receiving study medication.
Measure: Number; unit: Participants
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Participants | 9 | 11 | 8

4. Secondary Outcome: Time to Achieve First Confirmed Renal Improvement (RI) During Short-term Period (as Determined by Kaplan-Meier Methodology)
Description: RI is defined as meeting all of the following criteria. Renal function: If MDRD is abnormal at screening, within 10% of the MDRD at screening; if MDRD is 60-89 at screening, greater than or equal to 50% improvement based on the screening value or 90% or greater of MDRD at screening; if MDRD is 15-59 at screening, if MDRD is normal at screening-within 10% of the MDRD at screening. Proteinuria: improvement greater than or equal to 50% from screening. Hematuria: red blood cell (RBC)count within normal limit of central laboratory. Pyuria: white blood cell (WBC) count within normal limit of central laboratory. Cylindruria: No RBC or WBC casts.
Time Frame: Day 1 (randomization) to 12 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Abatacept 30/10 mg/kg: Abatacept 30/10 mg/kg regimen by IV infusion: abatacept 30 mg/kg on Days 1, 15, 29, and 57, followed by abatacept approximating 10 mg/kg on Days 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Days | 141 [88 to 169] | 136 [92 to 171] | 144 [113 to 198]
Statistical Analysis 1: Comparison: Abatacept 30/10 mg/kg vs Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 1.3, 95% CI 2-sided [0.91 to 1.78] — Point Estimate, 95% CI for the hazard ratio was determined by a Cox proportional hazards model including treatment as a covariate and stratified by prior treatment status
Statistical Analysis 2: Comparison: Abatacept 10/10 mg/kg vs Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 1.3, 95% CI 2-sided [0.91 to 1.77] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Participants Achieving Renal Improvement (RI) or CRR at Month 12 During Short-term Period
Description: CRR defined as meeting all of 5 criteria. RF: (Glomerular filtration rate [GFR] calculated using MDRD equation) Calculated function abnormal at screening visit - return of renal function to greater than or equal to 90% of function at approximately 6 months prior to onset of the current episode of lupus nephritis. Calculated function normal at screening visit - estimated renal function 90% or greater of level at screening visit. Proteinuria: urinary protein/creatinine ratio <30 mg/mmol. Hematuria: red blood cell (RBC) count within normal limits of Central Laboratory. Pyuria: White blood cell count (WBC) within normal limits of Central Laboratory. Cylindruria: No RBC or WBC casts reported.
Time Frame: At Month 12 from Day 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Participants | 38 [28.8 to 48.0] | 37 [27.8 to 46.9] | 31 [21.9 to 40.1]

6. Secondary Outcome: Number of Months CRR Was Maintained During Short-term Period
Description: Durability of CRR, defined as the number of months (number of consecutive planned visits beyond Day 15) a participant met the definition of CRR during the double-blind treatment period. Refer to outcome 1 for description of CRR.
Time Frame: Day 1 (randomization) to 12 Months
Population: All randomized participants who received participants.
Measure: Median (Full Range); unit: Months
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Months | 0 (1.5) [0 to 11] | 0 (1) [0 to 8] | 0 (1.1) [0 to 11]

7. Secondary Outcome: Baseline Renal Function Over Time During Short-term Period
Description: Baseline (BL) renal function, as estimated by calculation of the MDRD (Modification of Diet in Renal Disease) equation, over time. Renal MDRD is an equation (calculation) used to estimate Glomerular Filtration Rate (GFR) in participants with impaired renal function based on serum creatinine, age, race, and gender. GFR (mL/min/1.73 m^2) = 175 * (Scr)^-1.154 * (Age)^-0.203 * (0.742 if female) * (1.212 if African American) (conventional units). mL, milliliters; min, minute; m^2, meters squared; Scr, serum creatinine. A negative value indicates worsening.
Time Frame: Baseline (Day 1), Day 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, 337, 365
Population: n= Number of participants with measurements for that time point. Time-matched baseline (Day 1) values and post-baseline values are presented for each post-baseline visit and represent only that cohort of participants with measurement available at that post-baseline assessment.
Measure: Mean (Standard Deviation); unit: milliliters per minute (mL/min)/1.73 m^2
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
milliliters per minute (mL/min)/1.73 m^2
  Baseline (Day 1) for Day 15 (n=98,94,98) | 92.57 (36.57) | 99.09 (35.41) | 91.01 (29.60)
  Baseline (Day 1) for Day 29 (n=98,95,98) | 93.08 (36.14) | 98.56 (36.26) | 91.23 (29.33)
  Baseline (Day 1) for Day 57 (n=94, 89, 96) | 91.54 (35.99) | 98.76 (35.96) | 91.58 (28.93)
  Baseline (Day 1) for Day 85 (n=90, 91, 93) | 94.53 (35.53) | 100.22 (35.50) | 92.76 (29.01)
  Baseline (Day 1) for Day 113 (n=91, 83, 91) | 94.43 (35.80) | 101.23 (35.38) | 92.41 (28.15)
  Baseline (Day 1) for Day 141 (n=89, 83, 90) | 93.62 (35.74) | 101.05 (35.73) | 92.83 (29.10)
  Baseline (Day 1) for Day 169 (n=83, 82, 85) | 94.83 (36.10) | 101.95 (35.82) | 92.56 (29.85)
  Baseline (Day 1) for Day 197 (n=84, 81, 87) | 94.55 (35.98) | 101.85 (36.26) | 92.69 (29.51)
  Baseline (Day 1) for Day 225 (n=84, 81, 84) | 94.87 (35.82) | 101.64 (36.26) | 93.25 (29.75)
  Baseline (Day 1) for Day 253 (n=81, 76, 81) | 94.89 (36.24) | 101.25 (36.67) | 93.38 (30.07)
  Baseline (Day 1) for Day 281 (n=78, 77, 80) | 94.17 (36.55) | 102.64 (36.76) | 93.13 (30.13)
  Baseline (Day 1) for Day 309 (n=77, 76, 78) | 94.74 (36.81) | 100.64 (33.80) | 92.71 (30.23)
  Baseline (Day 1) for Day 337 (n=74, 75, 79) | 95.51 (37.30) | 101.00 (33.89) | 92.90 (30.13)
  Baseline (Day 1) for Day 365 (n=75, 73, 78) | 95.04 (37.24) | 101.30 (34.21) | 93.03 (30.53)

8. Secondary Outcome: Change in Renal Function From Baseline Over Time During Short-term Period
Description: Mean change from baseline in renal function, as estimated by calculation of the MDRD equation, over time. Renal MDRD is an equation (calculation) used to estimate Glomerular Filtration Rate (GFR) in participants with impaired renal function based on serum creatinine, age, race, and gender. GFR (mL/min/1.73 m^2) = 175 * (Scr)^-1.154 * (Age)^-0.203 * (0.742 if female) * (1.212 if African American) (conventional units). mL, milliliters; min, minute; m^2, meters squared; Scr, serum creatinine. A positive value indicates improvement. Change from baseline=Post-baseline-baseline value.
Time Frame: Baseline (Day 1), Day 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, 337, 365
Population: ITT population (all randomized and treated subjects). n= Number of participants with both baseline and post-baseline measurements for that time point.
Measure: Mean (Standard Error); unit: milliliters per minute (mL/min)/1.73 m^2
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
milliliters per minute (mL/min)/1.73 m^2
  Day 15; (n=98,94,98) | -0.24 (2.08) | 1.15 (2.11) | 0.62 (1.41)
  Day 29 (n=98, 95, 98) | 2.26 (1.87) | 4.51 (2.60) | 1.70 (1.88)
  Day 57 (n=94 89 96) | 5.96 (2.13) | 7.28 (3.38) | 2.38 (2.27)
  Day 85 (n=90, 91, 93) | 8.56 (2.88) | 6.20 (3.30) | 2.89 (2.30)
  Day 113 (n=91, 83, 91) | 5.31 (2.73) | 10.23 (4.11) | 4.12 (2.70)
  Day 141 (n=89, 83, 90) | 8.33 (2.74) | 7.90 (3.00) | 3.62 (2.28)
  Day 169 (n=83, 82, 85) | 8.12 (2.70) | 10.55 (3.46) | 7.34 (2.31)
  Day 197 (n=84, 81, 87) | 7.71 (2.73) | 10.67 (2.78) | 6.79 (2.25)
  Day 225 (n=84, 81, 84) | 7.32 (2.78) | 7.72 (2.77) | 7.19 (2.23)
  Day 253 (n=81, 76, 81) | 4.70 (3.02) | 7.22 (3.50) | 5.86 (2.39)
  Day 281 (n=78, 77, 80) | 5.68 (2.83) | 6.81 (3.37) | 5.38 (2.30)
  Day 309 (n=77, 76, 78) | 6.34 (2.89) | 9.53 (2.95) | 6.00 (2.57)
  Day 337 (n=74, 75, 79) | 5.34 (2.60) | 10.15 (2.74) | 4.39 (2.86)
  Day 365 (n=75, 73, 78) | 5.17 (2.75) | 11.03 (2.85) | 5.68 (2.49)

9. Secondary Outcome: Baseline and Post Baseline Systemic Lupus International Collaborating Clinics (SLICC)/American College of Rheumatology (ACR) Damage Index During Short-term Period
Description: SLICC/ACR score or damage index is a measure of cumulative damage due to Systemic Lupus Erythematosus (SLE). Damage is defined as nonreversible change (not related to active inflammation) occurring since onset of lupus, ascertained by clinical assessment and present for at least 6 months. A score of 0=no damage, early damage is defined as ≥1. The total maximum score is 48, and increasing score indicates increasing disease severity.
Time Frame: Baseline (Day 1), Post baseline (Month 12 or 28 days after last dose)
Population: n=Participants with both post-baseline and baseline measurements showing non-reversible changes in the SLICC/ACR Damage Index (i.e., Change from Baseline greater than or equal to 0).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Units on a scale
  Baseline (n=68, 67, 70) | 0.34 (0.68) | 0.27 (0.62) | 0.29 (0.73)
  Post Baseline Mean (n=68, 67, 70) | 0.53 (1.04) | 0.40 (0.80) | 0.44 (0.81)

10. Other Pre Specified Outcome: Number of Participants Achieving Patient Response (PR) at Month 12 During the Short-term Period
Description: PR is either CRR, Partial Renal Response(PRR),or no Response(NR).
  CRR= Serum creatinine(SC)is normal, Inactive urinary sediment, No cellular casts, Urinary protein/creatinine (UPCR) ratio <56.5 mg/mmoL; PRR= SC is normal OR SC not >25% above BL, RBCs at reference range, UPCR <56.5 mg/mmoL OR ≥50% improvement in UPCR with one of the following: UPCR <113 or <339 mg/mmoL, based on the BL ratio; NR= Not achieving either a CRR or a PRR. Participants achieved response if criteria at both months 11 and 12 (Days 337 and 365) were met. Participants who Early discontinuations were categorized as NR.
Time Frame: Month 12
Population: All randomized participants who received treatment.
Measure: Number; unit: Participants
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Participants
  No Renal Response | 61 | 69 | 66
  Partial Renal Response | 14 | 9 | 14
  Complete Renal Response | 24 | 21 | 20
Statistical Analysis 1: Comparison: Abatacept 30/10 mg/kg vs Placebo; Test type: Superiority or Other; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.68 to 21.3]
Statistical Analysis 2: Comparison: Abatacept 10/10 mg/kg vs Placebo; Test type: Superiority or Other; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.49 to 1.59]

11. Secondary Outcome: Number of Participants Achieving Renal Response (RR) at Month 12 During Short-term Period
Description: RR is defined as meeting BOTH of the following criteria:RENAL FUNCTION: Less than or equal to 25% increase from baseline;PROTEINURIA: Greater than or equal to 50% improvement in the urine protein/creatinine ratio with one of the following - urine protein/creatinine ratio (UPCR) <113 mg/mmol,, if the baseline ratio was <=339 mg/mmol OR UPCR <339 mg/mmol,if the baseline ratio > 339 mg/mmol. A participant was considered as achieving RR if response criteria at both months 11 and 12 (Days 337 and 365, respectively) were met. For 95% CI within each group, normal approximation is used if n>=5.
Time Frame: Month 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Participants | 45 [35.6 to 55.3] | 39 [29.8 to 49.0] | 33 [23.8 to 42.2]

12. Secondary Outcome: Change in SLICC/ACR Damage Index From Baseline During Short-term Period
Description: SLICC/ACR score or damage index is a measure of cumulative damage due to Systemic Lupus Erythematosus (SLE). Damage is defined as non-reversible change (not related to active inflammation) occurring since onset of lupus, ascertained by clinical assessment and present for at least 6 months. A score of 0=no damage, early damage is defined as ≥1. The total maximum score is 48, and increasing score indicates increasing disease severity. Change from baseline=Postbaseline - baseline value.
Time Frame: Baseline (Day 1), Postbaseline (Month 12 or 28 days after last dose)
Population: All randomized participants who received treatment and who had postbaseline and baseline measurements showing nonreversible changes (change from baseline >=0) in the SLICC-ACR Damage Index
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 68 | 67 | 70
Units on a scale | 0.17 (0.06) | 0.11 (0.06) | 0.13 (0.06)
Statistical Analysis 1: Comparison: Abatacept 30/10 mg/kg vs Placebo; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.13 to 0.19] — Adjustment based on ANCOVA model with treatment as factor and randomization strata (prior treatment status) and baseline measurements as covariates
Statistical Analysis 2: Comparison: Abatacept 10/10 mg/kg vs Placebo; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.18 to 0.14] — [estimate comment as in outcome 12, analysis 1]

13. Secondary Outcome: Baseline Physical Component Summary of the Short Form (SF)-36 During Short-term Period
Description: The SF-36 is a validated instrument measuring health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores (1) physical component summary=physical functioning, role-physical, bodily pain, and general health; (2) mental component summary=vitality, social functioning, role-emotional, and mental health. There is no total overall score; scoring is done for both subscores and summary scores. For subscores and summary scores, 0 =worst score (or quality of life) and 100=best score. Change from Baseline= post-Baseline - Baseline value.
Time Frame: Baseline (Day 1), Days 85, 169, 253, and 365
Population: n= Number of participants with both post-baseline and baseline measurements. Time-matched baseline (Day 1) values and post-baseline values are presented for each post-baseline visit and represent only that cohort of participants with measurement available at that post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Units on a scale
  Baseline (Day 1) for Day 85 (n=89, 91, 93) | 42.18 (9.07) | 43.80 (8.42) | 42.68 (8.93)
  Baseline (Day 1) for Day 169 (n=92, 94, 96) | 42.04 (9.08) | 44.17 (8.55) | 42.48 (8.90)
  Baseline (Day 1) for Day 253 (n=92, 94, 96) | 42.04 (9.08) | 44.17 (8.55) | 42.48 (8.90)
  Baseline (Day 1) for Day 365 (n=92, 94, 96) | 42.04 (9.08) | 44.17 (8.55) | 42.48 (8.90)

14. Secondary Outcome: Change From Baseline in Physical Component Summary of the SF-36 During Short-term Period
Description: as for outcome 13
Time Frame: Baseline (Day 1), Days 85, 169, 253, and 365
Population: ITT population; all randomized and treated subjects. To be included in analysis of change from baseline to time point with last observation carried forward, subjects must have had a baseline measurement and at least 1 post baseline measurement. n= Number of participants with both post-baseline and baseline measurements.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Units on a scale
  Day 85 (n=89, 91, 93) | 4.17 (0.82) | 2.61 (0.81) | 2.86 (0.80)
  Day 169 (n=92, 94, 96) | 4.18 (0.85) | 4.07 (0.84) | 3.39 (0.83)
  Day 253 (n=92, 94, 96) | 4.23 (0.92) | 4.80 (0.91) | 3.45 (0.90)
  Day 365 (n=92, 94, 96) | 4.24 (0.91) | 5.00 (0.91) | 3.77 (0.90)

15. Secondary Outcome: Baseline Mental Component Summary of the Short SF-36 During Short-term Period
Description: as for outcome 13
Time Frame: Baseline (Day 1), Days 85, 169, 253, and 365
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Units on a scale
  Baseline (Day 1) for Day 85 ( n=89, 91, 93) | 42.18 (9.07) | 43.80 (8.42) | 42.68 (8.93)
  Baseline (Day 1) for Day 169 (n=92,94,96) | 44.08 (10.93) | 41.84 (11.50) | 42.59 (12.22)
  Baseline (Day 1) for Day 253 ( n=92,94,96) | 44.08 (10.93) | 41.84 (11.50) | 42.59 (12.22)
  Baseline (Day 1) for Day 365 ( n=92,94,96) | 44.08 (10.93) | 41.84 (11.50) | 42.59 (12.22)

16. Secondary Outcome: Change From Baseline in Mental Component Summary of the SF-36 During Short-term Period
Description: as for outcome 13
Time Frame: Baseline (Day 1), Days 85, 169, 253, and 365
Population: ITT population; all randomized and treated subjects. To be included in analysis of change from baseline to time point with last observation carried forward (LOCF), participants must have had a baseline measurement and at least 1 post baseline measurement. n= Number of participants with both post-baseline and baseline measurements.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Units on a scale
  Day 85 (n=89, 91, 93) | 1.07 (1.11) | 3.10 (1.08) | 1.87 (1.08)
  Day 169 (n=92, 94, 96) | 2.90 (1.01) | 5.08 (1.00) | 3.69 (0.99)
  Day 253 (n=92, 94, 96) | 2.45 (1.00) | 4.83 (0.99) | 2.99 (0.98)
  Day 365 (n=92, 94, 96) | 2.62 (0.96) | 4.23 (0.95) | 2.84 (0.94)

17. Secondary Outcome: Baseline Fatigue as Measured by the Fatigue Visual Analog Scale During Short-term Period
Description: A visual analogue scale (VAS) is a psychometric response scale for measurement of subjective characteristics or attitudes that cannot be directly measured. The VAS for Fatigue (VAS-F) consists of a 100 mm line, with 0 (No Fatigue) on 1 end and 100 (Extreme Fatigue) on the other end, which a participant marks to indicate how much fatigue he or she feels. The marked point in mm is converted into a numeric value from 0 to 100, where 0=no fatigue and 100=maximum fatigue. Increasing numbers=increasing fatigue.
Time Frame: Baseline (Day 1), Days 85, 169, 253, and 365
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Units on a scale
  Baseline (Day 1) for Day 85 (n=90, 94, 95) | 48.86 (25.97) | 41.95 (22.81) | 48.93 (25.47)
  Baseline (Day 1) for Day 169 (n=92, 94, 97) | 48.80 (25.96) | 41.95 (22.81) | 48.25 (25.68)
  Baseline (Day 1) for Day 253 (n=92, 94, 97) | 48.80 (25.96) | 41.95 (22.81) | 48.25 (25.68)
  Baseline (Day 1) for Day 365 (n=92, 94, 97) | 48.80 (25.96) | 41.95 (22.81) | 48.25 (25.68)

18. Secondary Outcome: Change in Fatigue From Baseline as Measured by the Fatigue Visual Analog Scale During Short-term Period
Description: A visual analogue scale is a psychometric response scale for measurement of subjective characteristics or attitudes that cannot be directly measured.
  The VAS for Fatigue (VAS-F) consists of a 100 mm line, with 0 (No Fatigue) on 1 end and 100 (Extreme Fatigue) on the other end, which a participant marks to indicate how much fatigue he or she feels. The marked point in mm is converted into a numeric value from 0 to 100, where 0=no fatigue and 100=maximum fatigue. Increasing numbers=increasing fatigue.
Time Frame: Baseline (Day 1), Days 85, 169, 253, and 365
Population: ITT population; all randomized and treated subjects. To be included in analysis of change from baseline to time point with last observation carried forward, participants must have had a baseline measurement and at least 1 post baseline measurement. n= Number of participants with both post-baseline and baseline measurements.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Units on a scale
  Day 85 (n=90, 94, 95) | -9.18 (2.37) | -4.94 (2.33) | -6.20 (2.33)
  Day 169 (n=92, 94, 97) | -7.18 (2.49) | -9.52 (2.48) | -4.71 (2.44)
  Day 253 (n=92, 94, 97) | -8.78 (2.59) | -11.90 (2.57) | -7.35 (2.53)
  Day 365 (n=92, 94, 97) | -12.21 (2.70) | -12.32 (2.69) | -11.07 (2.65)

19. Secondary Outcome: Baseline Fatigue as Measured by Fatigue Severity Scale-Krupp During Short-term Period
Description: The reduction of fatigue assessed by Fatigue Severity Scale (FSS). The FSS questionnaire is comprised of 9 statements inquiring about the examinee's sleep habits over the preceding week. Participants are asked to rate their level of agreement (toward seven) or disagreement (toward zero) with the nine statements. A score of 36 and above (out of a maximum of 63) indicates the presence of significant fatigue.
Time Frame: Baseline (Day 1), Days 85, 169, 253, and 365
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Units on a scale
  Baseline (Day 1) for Day 85 (n=90, 94, 95) | 40.60 (13.75) | 39.14 (13.54) | 39.64 (13.00)
  Baseline (Day 1) for Day 169 (n=92, 94, 97) | 40.41 (13.67) | 39.14 (13.54) | 39.59 (12.87)
  Baseline (Day 1) for Day 253 ( n=92, 94, 97) | 40.41 (13.67) | 39.14 (13.54) | 39.59 (12.87)
  Baseline (Day 1) for Day 365 ( n=92, 94, 97) | 40.41 (13.67) | 39.14 (13.54) | 39.59 (12.87)

20. Secondary Outcome: Change in Fatigue From Baseline as Measured by Fatigue Severity Scale-Krupp During Short-term Period
Description: as for outcome 19
Time Frame: Baseline (Day 1), Days 85, 169, 253, and 365
Population: ITT population (all randomized and treated subjects). To be included in analysis of change from baseline to time point with last observation carried forward, subjects must have had a baseline measurement and at least 1 post baseline measurement. n= Number of participants with both post-baseline and baseline measurements.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Units on a scale
  Day 85 (n=90, 94, 95) | -1.54 (1.20) | -1.40 (1.18) | -0.67 (1.18)
  Day 169 (n=92, 94, 97) | -2.68 (1.15) | -1.69 (1.14) | -1.08 (1.13)
  Day 253 ( n=92, 94, 97) | -3.54 (1.12) | -2.95 (1.11) | -3.06 (1.09)
  Day 365 ( n=92, 94, 97) | -4.20 (1.21) | -3.21 (1.20) | -4.79 (1.19)

21. Secondary Outcome: Participants With Adverse Events (AEs), Serious AEs (SAEs), Deaths, and Discontinuations Due to AEs Reported During the Short-term Period
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=possibly, probably, or certainly related to and of unknown relationship to study drug.
Time Frame: From Baseline (Day 1) up to 56 days post last dose in the double-blind period or the first dose in the open-label long-term extension, whichever occurred first.
Population: All participants who received at least one dose of double-blind study medication were included in the safety population.
Measure: Number; unit: Participants
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Participants
  Deaths | 5 | 2 | 7
  SAEs | 33 | 28 | 31
  Related SAEs | 20 | 19 | 15
  AEs | 93 | 89 | 94
  Related AEs | 61 | 53 | 55
  Discontinued due to AEs | 14 | 13 | 9

22. Secondary Outcome: Participants With AEs of Special Interest During the Short-term Period
Description: AEs of special interest were prospectively identified to be those that may be associated with the use of immunomodulatory agents. They are a subset of all AEs and may be either serious or non-serious.
Time Frame: as for outcome 21
Population: All participants who received at least one dose of double-blind study medication were included in the safety population.
Measure: Number; unit: Participants
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Participants
  Infections and Infestations | 75 | 70 | 75
  Malignancies | 0 | 1 | 1
  Autoimmune Disorders | 4 | 5 | 3
  Acute Infusional AEs | 23 | 18 | 17
  Peri-infusional AEs | 23 | 18 | 17

23. Secondary Outcome: Participants With Marked Hematology Abnormalities During the Short-term Period
Description: LLN=lower limit of normal; ULN=upper limit of normal; PTV=pretreatment value. Normal ranges are provided by the Central Laboratory and may vary according to sex and age. Low(↓)Hemoglobin:>3g/dL decrease from PTV; ↓Hematocrit:<0.75xPTV;↓Erythrocyte count:<0.75xPTV; high(↑)Platelet count:>1.5xULN;↓Platelet count:<0.67xLLN;↓Leukocyte count:<0.75X LLN;↑Leukocyte count:>1.25xULN;↓Absolute(AB)Neutrophils+Bands:<1.00x10^3c/uL;↑AB Lymphocyte count:>7.50x10^3 c/uL; ↓AB lymphocyte count:<0.750x10^3 c/uL;↑AB monocyte count:>2000/mm^3;↑AB basophil count:>400/mm^3;↑AB eosinophil count:>0.750x10^3 c/uL.
Time Frame: as for outcome 21
Population: All participants who received at least one dose of double-blind study medication were included in the safety population. n= number of participants with both post-baseline and baseline measurements
Measure: Number; unit: Participants
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Participants
  Low Hemoglobin (n=98, 98, 99) | 6 | 3 | 9
  Low Hematocrit (n=97, 98, 99) | 5 | 1 | 7
  Low Erythrocyte Count (n=98, 98, 99) | 4 | 1 | 7
  High Platelet Count (n=98, 98, 98) | 1 | 0 | 1
  Low Platelet Count (n=98, 98, 98) | 1 | 3 | 1
  High Leukocyte Count (n=98, 98, 99) | 15 | 10 | 11
  Low Leukocyte Count (n=98,98,99) | 13 | 18 | 16
  Low Absolute Neutrophils + Bands (n=98,98,99) | 1 | 2 | 7
  High Absolute Lymphocyte Count (n=98,98,99) | 0 | 2 | 0
  Low Absolute Lymphocyte Count (n=98, 98, 99) | 47 | 32 | 53
  High Absolute Monocyte Count (n=98, 98, 99) | 1 | 1 | 1
  High Absolute Basophil Count (n=98, 98, 99) | 0 | 0 | 0
  High Absolute Eosinophil Count (n=98, 98, 99) | 0 | 3 | 0

24. Secondary Outcome: Participants With Marked Laboratory Abnormalities During the Short-term Period
Description: LLN=lower limit of normal; ULN=upper limit of normal; PTV=pretreatment value. Normal ranges are provided by the Central Laboratory and may vary according to sex and age. ↑Serum Sodium:>1.05x ULN;↓Serum Potassium:<0.9x LLN;↑Serum Potassium:>1.1x ULN;↓Total Calcium:<0.8X LLN;↑Total Calcium:>1.2x ULN; ↓Serum Glucose(SG):<65 mg/dL;↑SG:>220 mg/dL;↓Fasting SG:<0.8x LLN;↑Fasting SG:>1.5x ULN;↓Total Protein:<0.9x LLN;↓Albumin:<0.9x LLN;↑Total Cholesterol:>2x PTV;↑Triglycerides:>=2.5x ULN;↑Fasting Triglycerides:>=2x ULN
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Participants
  High Serum Sodium (n=98, 98, 99) | 1 | 2 | 0
  Low Serum Potassium (n=98, 98, 99) | 12 | 14 | 15
  High Serum Potassium (n=98, 98, 99) | 4 | 0 | 2
  Low Total Calcium (n=98, 98, 99) | 0 | 1 | 1
  High Total Calcium (n=98, 98, 99) | 1 | 2 | 1
  Low Serum Glucose (n=98, 98, 99) | 12 | 16 | 18
  High Serum Glucose (n=98, 98, 99) | 2 | 2 | 2
  Low Fasting Serum Glucose (n=72, 73, 68) | 3 | 2 | 0
  High Fasting Serum Glucose (n=72, 73, 68) | 1 | 1 | 0
  Low Total Protein (n=98, 98, 99) | 18 | 18 | 25
  Low Albumin (n=98, 98, 99) | 10 | 6 | 4
  High Total Cholesterol (n=93,93,96) | 2 | 0 | 1
  High Triglycerides (n=71, 79, 75) | 2 | 0 | 0
  High Fasting Triglycerides (n=65, 64, 63) | 3 | 0 | 0

25. Secondary Outcome: Participants With Marked Liver and Kidney Function Abnormalities During the Short-term Period
Description: ULN=upper limit of normal; PTV=pretreatment value. Normal ranges are provided by the Central Laboratory and may vary according to sex and age.
  Alkaline Phosphatase:>2x ULN; ↑Aspartate Aminotransferase: >3x ULN; ↑Alanine Aminotransferase : >3x ULN; G-Glutamyl Transferase : >2x ULN; ↑Total Bilirubin : >2x ULN or if PTV > ULN then > 4x PTV; ↑Blood Urea Nitrogen >2x PTV; ↑Creatinine >1.5x PTV.
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
Participants
  High Alkaline Phosphatase | 1 | 1 | 1
  High Aspartate Aminotransferase | 2 | 0 | 0
  High Alanine Aminotransferase | 7 | 4 | 1
  High G-Glutamyl Transferase | 7 | 7 | 5
  High Total Bilirubin | 0 | 0 | 0
  High Blood Urea Nitrogen | 5 | 1 | 6
  High Creatinine | 16 | 6 | 12

26. Secondary Outcome: Participants With Marked Abnormalities Urinalysis During the Short-term Period
Description: PTV=pretreatment value. Criteria for marked abnormality: Protein, glucose, blood, leukocyte esterase , if missing PTV then use >=2+ (or, if value >=4, or if PTV=0 or 0.5, >=2 or if PTV=1, >=3, or if PTV=2 or 3, >=4).
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 98 | 99
Participants
  Urine Protein (n=99,98,99) | 6 | 3 | 8
  Urine Glucose (n=99,98,99) | 1 | 3 | 0
  Urine Blood (n=99,98,99) | 16 | 19 | 17
  Urine Leukocyte esterase (n=85,91,90) | 10 | 8 | 8

27. Secondary Outcome: Vital Signs Summary During the Short-term Period: Systolic Blood Pressure (SBP)
Time Frame: 0 - 12 Months
Population: All participants who received at least one dose of double-blind study medication were included in the safety population. n= number of participants with a measurement at the select time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
mmHg
  Day 1: SBP-before infusion; n=76,81,73 | 128.2 (16.34) | 127.8 (15.86) | 126.2 (16.88)
  Day 1: SBP-1hour after infusion; n=69,78,70 | 127.7 (17.60) | 126.7 (15.53) | 126.0 (18.20)
  Day 1: SBP-2.5 hours after infusion; n=79,81,76 | 127.1 (16.92) | 127.8 (12.55) | 126.2 (15.82)
  Day 15: SBP-before infusion; n=78,78,74 | 127.6 (18.71) | 125.5 (16.42) | 129.2 (17.80)
  Day 15: SBP- 1hour after infusion; n=72,75,71 | 126.9 (14.79) | 125.9 (16.35) | 128.2 (14.65)
  Day 15: SBP-2.5 hours after infusion; n=80,78,78 | 130.1 (14.99) | 124.9 (15.08) | 131.2 (15.58)
  Day 29: SBP-before infusion; n=77,79,75 | 125.6 (13.52) | 126.2 (15.31) | 126.9 (14.79)
  Day 29: SBP-1hour after infusion; n=72,75,74 | 126.2 (12.92) | 125.9 (15.85) | 128.6 (15.34)
  Day 29: SBP-2.5 hours after infusion; n=80,79,82 | 126.3 (13.77) | 126.4 (14.86) | 127.6 (14.54)
  Day 57: SBP-before infusion; n=74,76,70 | 126.4 (15.47) | 124.8 (16.21) | 123.0 (13.21)
  Day 57: SBP-1hour after infusion; n=74,69,68 | 124.6 (13.40) | 122.1 (16.73) | 124.4 (11.22)
  Day 57: SBP-2.5 hours after infusion; n=81,73,73 | 127.0 (13.04) | 123.6 (14.43) | 126.1 (14.29)
  Day 85: SBP- before infusion; n=73,71,67 | 122.0 (13.52) | 118.7 (12.85) | 122.2 (13.67)
  Day 85: SBP-1hour after infusion; n=73,69,72 | 121.8 (13.28) | 119.6 (13.59) | 122.0 (14.23)
  Day 113: SBP-before infusion; n=72,70,70 | 122.6 (18.07) | 121.7 (14.26) | 119.9 (14.16)
  Day 113: SBP-1hour after infusion; n=75,70,75 | 121.5 (16.81) | 121.0 (13.13) | 120.1 (14.69)
  Day 141: SBP-before infusion; n=66,70,66 | 121.4 (15.94) | 119.2 (15.67) | 118.8 (14.26)
  Day 141: SBP-1hour after infusion; n=72,71,70 | 120.9 (18.11) | 117.9 (15.32) | 120.4 (13.26)
  Day 169: SBP-before infusion; n=70,70,66 | 118.5 (16.30) | 117.6 (12.13) | 118.6 (14.65)
  Day 169: SBP-1hour after infusion; n=75,71,71 | 120.3 (18.74) | 118.2 (11.83) | 118.9 (14.15)
  Day 197: SBP-before infusion; n=68,70,64 | 119.0 (15.58) | 118.9 (14.72) | 118.7 (12.34)
  Day 197: SBP-1hour after infusion; n=72,73,70 | 117.7 (14.76) | 117.4 (13.10) | 120.4 (15.29)
  Day 225: SBP-before infusion; n=70,64,63 | 118.2 (14.53) | 118.8 (13.51) | 119.5 (13.20)
  Day 225: SBP-1hour after infusion; n=72,65,68 | 116.6 (15.82) | 119.5 (14.60) | 118.8 (12.83)
  Day 253: SBP-before infusion; n=63,66,63 | 120.6 (15.13) | 120.2 (17.21) | 120.9 (14.17)
  Day 253: SBP-1hour after infusion; n=69,67,67 | 118.1 (14.81) | 117.1 (15.02) | 119.7 (14.16)
  Day 281: SBP-before infusion; n=63,66,58 | 120.7 (14.02) | 116.5 (14.30) | 120.3 (12.78)
  Day 281: SBP-1hour after infusion; n=66,65,64 | 119.5 (15.28) | 119.4 (13.70) | 121.0 (12.48)
  Day 309: SBP-before infusion; n=63,63,59 | 119.4 (14.18) | 116.3 (14.33) | 120.5 (15.32)
  Day 309: SBP-1hour after infusion; n=67,66,64 | 119.6 (13.47) | 114.1 (14.97) | 119.2 (15.73)
  Day 337: SBP-before infusion; n=63,64,61 | 119.9 (12.52) | 117.3 (14.71) | 119.3 (14.49)
  Day 337: SBP-1hour after infusion; n=68,65,67 | 120.4 (12.97) | 117.7 (16.48) | 119.3 (13.67)

28. Secondary Outcome: Vital Signs Summary During the Short-term Period: Diastolic Blood Pressure (DBP)
Time Frame: 0 - 12 Months
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 98 | 99
mm Hg
  Day 1: DBP-before infusion; n=76,81,73 | 80.8 (11.69) | 80.6 (12.57) | 80.4 (12.40)
  Day 1: DBP-1hour after infusion; n=69,78,70 | 79.6 (13.57) | 79.6 (12.59) | 80.1 (13.34)
  Day 1: DBP-2.5 hours after infusion; n=79,81,76 | 79.3 (12.73) | 79.0 (10.93) | 80.9 (11.24)
  Day 15: DBP-before infusion; n=78,78,74 | 81.1 (12.56) | 80.0 (12.89) | 82.6 (12.89)
  Day 15: DBP- 1hour after infusion; n=72,75,71 | 79.6 (10.87) | 78.7 (11.58) | 80.4 (10.96)
  Day 15: DBP-2.5 hours after infusion; n=80,78,78 | 81.4 (11.79) | 78.0 (11.27) | 82.8 (11.38)
  Day 29: DBP-before infusion; n=77,79,75 | 79.6 (11.08) | 78.8 (12.14) | 81.3 (9.95)
  Day 29: DBP-1hour after infusion; n=72,75,74 | 79.9 (10.06) | 78.0 (12.84) | 80.8 (10.36)
  Day 29: DBP-2.5 hours after infusion; n=80,79,82 | 78.5 (9.75) | 78.2 (11.62) | 79.5 (11.08)
  Day 57: DBP-before infusion; n=74,76,70 | 80.0 (10.98) | 78.7 (10.69) | 78.7 (10.59)
  Day 57: DBP-1hour after infusion; n=74,69,68 | 78.9 (11.23) | 75.3 (11.87) | 78.7 (9.25)
  Day 57: DBP-2.5 hours after infusion; n=81,73,73 | 79.5 (10.06) | 76.1 (10.49) | 80.2 (9.60)
  Day 85: DBP- before infusion; n=73,71,67 | 79.7 (11.01) | 75.2 (9.39) | 78.7 (9.94)
  Day 85: DBP-1hour after infusion; n=73,69,72 | 78.1 (11.72) | 75.6 (9.29) | 78.1 (10.58)
  Day 113: DBP-before infusion; n=72,70,70 | 78.5 (13.75) | 77.0 (10.58) | 76.7 (11.62)
  Day 113: DBP-1hour after infusion; n=75,70,75 | 76.1 (12.13) | 76.3 (10.74) | 76.9 (11.61)
  Day 141: DBP-before infusion; n=66,70,66 | 78.8 (11.32) | 74.0 (12.08) | 76.5 (11.48)
  Day 141: DBP-1hour after infusion; n=72,71,70 | 77.8 (11.24) | 74.7 (11.54) | 76.1 (11.69)
  Day 169: DBP-before infusion; n=70,70,66 | 75.5 (12.96) | 74.1 (10.18) | 77.0 (13.16)
  Day 169: DBP-1hour after infusion; n=75,71,71 | 76.5 (13.24) | 74.4 (9.41) | 76.4 (12.81)
  Day 197: DBP-before infusion; n=68,70,64 | 76.8 (11.29) | 75.8 (10.79) | 75.8 (11.16)
  Day 197: DBP-1hour after infusion; n=72,73,70 | 76.1 (11.63) | 74.5 (10.55) | 75.4 (12.21)
  Day 225: DBP-before infusion; n=70,64,63 | 74.5 (12.39) | 73.6 (9.68) | 75.7 (10.77)
  Day 225: DBP-1hour after infusion; n=72,65,68 | 75.0 (11.67) | 74.5 (10.95) | 76.0 (10.28)
  Day 253: DBP-before infusion; n=63,66,63 | 76.1 (11.54) | 75.9 (11.27) | 77.1 (10.26)
  Day 253: DBP-1hour after infusion; n=69,67,67 | 74.5 (11.51) | 74.9 (10.25) | 75.7 (10.20)
  Day 281: DBP-before infusion; n=63,66,58 | 77.6 (10.89) | 73.3 (9.50) | 76.6 (9.31)
  Day 281: DBP-1hour after infusion; n=66,65,64 | 75.9 (10.49) | 74.5 (9.73) | 76.6 (10.15)
  Day 309: DBP-before infusion; n=63,63,59 | 78.1 (9.73) | 72.9 (8.90) | 77.4 (11.83)
  Day 309: DBP-1hour after infusion; n=67,66,64 | 76.4 (10.81) | 72.9 (9.86) | 76.6 (10.75)
  Day 337: DBP-before infusion; n=63,64,61 | 78.0 (10.54) | 73.4 (9.52) | 76.2 (10.65)
  Day 337: DBP-1hour after infusion; n=68,65,67 | 78.1 (9.72) | 73.3 (9.82) | 76.1 (11.19)

29. Secondary Outcome: Vital Signs Summary During the Short-term Period: Heart Rate
Time Frame: 0 - 12 Months
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
beats per minute
  Day 1: before infusion; n=99,98,100 | 82.4 (11.17) | 79.2 (10.84) | 82.6 (12.11)
  Day 1: 1hour after infusion; n=98,98,98 | 81.3 (11.08) | 79.6 (9.71) | 81.9 (10.64)
  Day 1: 2.5 hours after infusion; n=97,96,96 | 81.8 (11.38) | 82.2 (11.25) | 83.8 (11.51)
  Day 15: before infusion; n=97,93,99 | 83.1 (12.08) | 81.0 (11.31) | 83.7 (12.84)
  Day 15: 1hour after infusion; n=96,94,98 | 81.3 (12.21) | 80.1 (11.31) | 82.6 (11.70)
  Day 15: 2.5 hours after infusion; n=93,92,95 | 81.5 (11.18) | 81.7 (9.88) | 84.7 (12.65)
  Day 29: before infusion; n=94,93,99 | 83.7 (12.13) | 80.8 (11.85) | 83.0 (12.91)
  Day 29: 1hour after infusion; n=93,92,99 | 81.7 (12.23) | 79.9 (9.60) | 81.7 (11.00)
  Day 29: 2.5 hours after infusion; n=92,90,97 | 81.3 (10.26) | 82.1 (9.56) | 84.7 (11.41)
  Day 57: before infusion; n=93,88,84 | 83.4 (11.04) | 82.2 (12.09) | 82.8 (13.00)
  Day 57: 1hour after infusion; n=93,84,94 | 81.0 (10.02) | 81.6 (10.52) | 81.8 (10.80)
  Day 57: 2.5 hours after infusion; n=91,84,91 | 82.5 (10.13) | 83.4 (12.20) | 83.8 (11.09)
  Day 85: before infusion; n=89,86,91 | 84.8 (12.35) | 82.3 (11.00) | 82.5 (10.99)
  Day 85: 1hour after infusion; n=88,84,89 | 83.3 (11.02) | 80.4 (10.67) | 83.5 (9.50)
  Day 113: before infusion; n=88,82,92 | 82.1 (11.46) | 80.4 (11.88) | 83.0 (11.78)
  Day 113: 1hour after infusion; n=87,80,91 | 81.8 (10.64) | 80.2 (9.98) | 82.6 (10.62)
  Day 141: before infusion; n=84,82,89 | 82.8 (11.75) | 79.3 (11.20) | 82.6 (12.74)
  Day 141: 1hour after infusion; n=84,81,86 | 81.4 (10.92) | 79.1 (10.59) | 81.3 (11.30)
  Day 169: before infusion; n=85,82,86 | 80.1 (10.01) | 78.0 (11.35) | 79.1 (10.95)
  Day 169: 1hour after infusion; n=84,82,85 | 79.5 (10.43) | 78.8 (10.97) | 81.4 (12.30)
  Day 197: before infusion; n=83,82,84 | 81.7 (10.54) | 78.1 (10.72) | 79.3 (11.58)
  Day 197: 1hour after infusion; n=82,82,85 | 79.8 (9.84) | 78.7 (10.25) | 79.6 (11.77)
  Day 225: before infusion; n=83,76,81 | 80.1 (10.04) | 77.6 (10.59) | 78.9 (10.00)
  Day 225: 1hour after infusion; n=83,76,81 | 79.1 (9.86) | 78.0 (9.83) | 80.2 (10.03)
  Day 253: before infusion; n=78,77,81 | 81.4 (11.32) | 79.1 (11.30) | 81.5 (12.17)
  Day 253: 1hour after infusion; n=78,77,81 | 78.8 (9.01) | 79.3 (10.64) | 79.5 (10.91)
  Day 281: before infusion; n=75,76,77 | 80.1 (10.56) | 78.3 (11.16) | 79.3 (10.24)
  Day 281: 1hour after infusion; n=74,76,76 | 78.0 (9.93) | 77.6 (9.46) | 78.7 (9.95)
  Day 309: before infusion; n=76,75,77 | 79.8 (10.89) | 76.5 (10.07) | 78.2 (10.66)
  Day 309: 1hour after infusion; n=76,74,77 | 77.9 (10.40) | 77.4 (9.81) | 78.4 (11.49)
  Day 337: before infusion; n=73,75,80 | 78.5 (11.77) | 76.4 (9.95) | 78.9 (11.50)
  Day 337: 1hour after infusion; n=73,73,79 | 77.6 (9.85) | 77.4 (9.73) | 78.3 (11.11)

30. Secondary Outcome: Vital Signs Summary During the Short-term Period: Temperature
Time Frame: 0 - 12 Months
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: degree celcius
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
degree celcius
  Day 1: before infusion; n=99,98,99 | 36.6 (0.48) | 36.5 (0.42) | 36.5 (0.47)
  Day 1: 1hour after infusion; n=98,96,97 | 36.6 (0.50) | 36.5 (0.46) | 36.6 (0.51)
  Day 1: 2.5 hours after infusion; n=97,93,97 | 36.6 (0.45) | 36.5 (0.43) | 36.6 (0.49)
  Day 15: before infusion; n=97,94,99 | 36.5 (0.50) | 36.5 (0.45) | 36.5 (0.47)
  Day 15: 1hour after infusion; n=96,91,98 | 36.6 (0.47) | 36.5 (0.45) | 36.5 (0.53)
  Day 15: 2.5 hours after infusion; n=93,91,95 | 36.6 (0.47) | 36.5 (0.44) | 36.6 (0.53)
  Day 29: before infusion; n=94,93,99 | 36.5 (0.51) | 36.4 (0.489) | 36.5 (0.48)
  Day 29: 1hour after infusion; n=93,91,98 | 36.5 (0.50) | 36.5 (0.44) | 36.5 (0.49)
  Day 29: 2.5 hours after infusion; n=92,90,97 | 36.5 (0.46) | 36.5 (0.47) | 36.5 (0.49)
  Day 57: before infusion; n=93,88,93 | 36.5 (0.46) | 36.4 (0.50) | 36.5 (0.49)
  Day 57: 1hour after infusion; n=93,83,94 | 36.1 (3.58) | 36.4 (0.46) | 36.6 (0.49)
  Day 57: 2.5 hours after infusion; n=90,84,90 | 36.5 (0.41) | 36.5 (0.48) | 36.5 (0.53)
  Day 85: before infusion; n=89,86,91 | 36.4 (0.52) | 36.4 (0.45) | 36.5 (0.45)
  Day 85: 1hour after infusion; n=87,84,89 | 36.4 (0.51) | 36.4 (0.50) | 36.5 (0.49)
  Day 113: before infusion; n=88,82,92 | 36.5 (0.60) | 36.4 (0.50) | 36.5 (0.54)
  Day 113: 1hour after infusion; n=87,79,91 | 36.4 (0.49) | 36.4 (0.44) | 36.5 (0.51)
  Day 141: before infusion; n=84,81,89 | 36.5 (0.50) | 36.4 (0.45) | 36.5 (0.47)
  Day 141: 1hour after infusion; n=84,80,86 | 36.5 (0.45) | 36.4 (0.41) | 36.5 (0.49)
  Day 169: before infusion; n=85,81,86 | 36.5 (0.52) | 36.4 (0.48) | 36.5 (0.46)
  Day 169: 1hour after infusion; n=84,80,84 | 36.4 (0.47) | 36.4 (0.44) | 36.5 (0.46)
  Day 197: before infusion; n=83,82,85 | 36.5 (0.58) | 36.3 (0.45) | 36.5 (0.45)
  Day 197: 1hour after infusion; n=82,81,84 | 36.4 (0.61) | 36.3 (0.49) | 36.5 (0.48)
  Day 225: before infusion; n=83,76,81 | 36.5 (0.56) | 36.4 (0.48) | 36.4 (0.55)
  Day 225: 1hour after infusion; n=83,75,81 | 36.5 (0.56) | 36.4 (0.45) | 36.5 (0.54)
  Day 253: before infusion; n=78,77,80 | 36.5 (0.52) | 36.4 (0.44) | 36.5 (0.46)
  Day 253: 1hour after infusion; n=78,77,81 | 36.5 (0.54) | 36.4 (0.42) | 36.5 (0.49)
  Day 281: before infusion; n=75,76,77 | 36.5 (0.49) | 36.4 (0.43) | 36.5 (0.49)
  Day 281: 1hour after infusion; n=74,76,76 | 36.5 (0.51) | 36.4 (0.46) | 36.5 (0.47)
  Day 309: before infusion; n=76,75,77 | 36.5 (0.49) | 36.3 (0.51) | 36.5 (0.54)
  Day 309: 1hour after infusion; n=75,73,77 | 36.5 (0.51) | 36.4 (0.43) | 36.5 (0.54)
  Day 337: before infusion; n=73,75,79 | 36.5 (0.47) | 36.4 (0.46) | 36.5 (0.50)
  Day 337: 1hour after infusion; n=73,72,79 | 36.5 (0.59) | 36.4 (0.49) | 36.5 (0.52)

31. Secondary Outcome: Number of Participants With Positive Abatacept-induced Responses (ECL Method) Over Time During the Short-term Period
Description: A validated, sensitive electrochemiluminescence (ECL) immunoassay based on Meso-Scale Discovery instrumentation was used to evaluate immunogenicity. The ECL assay differentiated between two antibody specificities: (1) the 'Ig and/or Junction (Jn) Region' and (2) 'CLTA4 and possibly Ig'. A sample was considered positive if it had a titer of 10 or greater and if immunodepletion was observed with abatacept with or without CTLA4-T.
Time Frame: Day 169, Day 365
Population: Immunogenicity analysis population consisted of participants who received at least 1 dose of abatacept and had at least 1 immunogenicity result available. n= number of participants who are evaluated
Measure: Number; unit: Participants
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 95 | 96 | 0
Participants
  CTLA4 and possibly Ig; Day 169 (n=90) | 2 | 1 |
  CTLA4 and possibly Ig; Day 365 (n=74) | 1 | 0 |
  CTLA4 and possibly Ig;Overall on TRT visits (n=90) | 3 | 1 |
  CTLA4 and possibly Ig; Overall Post visits (n=20) | 7 | 5 |
  CTLA4 and possibly Ig; Overall (n=96) | 9 | 6 |
  Ig/Jn region; Day 169 (n=90) | 0 | 0 |
  Ig/Jn region; Day 365 (n=78) | 1 | 0 |
  Ig/Jn region; Overall on TRT visits (n=90) | 1 | 0 |
  Ig/Jn region; Overall on Post visits (n=20) | 0 | 1 |
  Ig/Jn region; Overall (n=95) | 1 | 1 |

32. Secondary Outcome: Baseline Quantitative Immunoglobulins During the Short-term Period
Description: A quantitative immunoglobulins (Igs) test is used to detect abnormal levels of the three major classes of Igs (IgG, IgA, and IgM). Abnormal test results typically indicate that there is something affecting the immune system which requires further testing.
Time Frame: Baseline (Day 1)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
mg/dL
  Immunoglobulin IgA | 246.28 (99.55) | 218.04 (88.23) | 230.23 (107.34)
  Immunoglobulin IgG | 939.80 (423.66) | 864.12 (459.44) | 1013.17 (516.24)
  Immunoglobulin IgM | 100.96 (79.70) | 97.10 (55.18) | 98.49 (57.71)

33. Secondary Outcome: Change in Quantitative Immunoglobulin From Baseline During Short-term Period
Description: A quantitative immunoglobulin (Ig) test is used to detect abnormal levels of the 3 major classes of Ig (IgG, IgA, and IgM). Abnormal test results typically indicate that something is affecting the immune system and further testing is required.
  Please refer to Outcome 31 for the respective baseline values
Time Frame: Day 365
Population: All randomized participants who received treatment. n=Participants with both postbaseline and baseline measurements
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 99 | 99 | 100
mg/dL
  Ig A (n=76, 73, 78) | -32.83 (8.47) | -34.48 (6.87) | -26.51 (8.20)
  IgG (n=76, 73, 78) | 41.41 (47.17) | 27.21 (43.84) | 23.42 (49.07)
  IgM (n=76, 73, 78) | -17.76 (5.28) | -19.38 (4.76) | -20.62 (4.89)

34. Secondary Outcome: Number of Participants Achieving Complete Response by ACCESS Definition
Description: The Abatacept and Cyclophosphamide Combination Efficacy and Safety Study (ACCESS) defines complete response as a response meeting all of the following criteria: serum creatinine ≤upper limit of normal as defined by the central laboratory or ≤125% of the higher value at either screening or baseline; urine protein/creatinine ratio <50 mg/mmoL; and prednisone or prednisone-equivalent dose tapered to 10 mg per day.
Time Frame: End of short-term period (Day 365) to termination of the long-term extension period
Population: All participants who entered and received at least 1 dose of study medication during the long-term extension period
Measure: Number; unit: participants
Groups:
- Abatacept 30/10 mg/kg: Short-term period: Abatacept 30/10 mg/kg regimen by intravenous (IV) infusion: abatacept 30 mg/kg on Days 1, 15, 29, and 57, followed by abatacept approximating 10 mg/kg on Days 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral mycophenolate mofetil (MMF) and oral prednisone or prednisone-equivalent Long-term extension period:Participants received abatacept in a weight-tiered dose of approximately 10 mg/kg administered every 28 days by IV infusion in addition to oral MMF and oral prednisone or prednisone-equivalent.
- Abatacept 10/10 mg/kg: Abatacept 10/10 mg/kg regimen by IV infusion: abatacept approximating 10 mg/kg on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent Long-term extension period:Participants received abatacept in a weight-tiered dose of approximately 10 mg/kg administered every 28 days by IV infusion in addition to oral MMF and oral prednisone or prednisone-equivalent.
- Placebo: Placebo (Dextrose 5% in water [D5W]) or Normal Saline (NS) by IV infusion on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent Long-term extension period:Participants received abatacept in a weight-tiered dose of approximately 10 mg/kg administered every 28 days by IV infusion in addition to oral MMF and oral prednisone or prednisone-equivalent.
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 69 | 66 | 74
participants
  Day 365 | 29 | 30 | 25
  Day 645 (n=55, 56, 61) | 27 | 28 | 25

35. Secondary Outcome: Number of Participants Achieving Patient Response of Complete or Partial Response, Based on the June 2010 Food and Drug Administration Guidance Document for Lupus Nephritis
Description: Patient response=complete, partial, or no response. Complete response=serum creatinine (SCr) normal, inactive urinary sediment, no cellular casts, urinary protein/creatinine (UPCR) ratio<56.5 mg/mmol. Partial response=SCr normal or ≤25% above baseline value, RBCs at reference range, UPCR <56.5 mg/mmoL OR ≥50% improvement in UPCR with one of the following: UPCR <113 or <339 mg/mmoL, based on the baseline ratio. No response=Not achieving complete or partial response criteria.
Time Frame: At Day 365 (end of Short-term Period) and Day 645
Population: All participants who entered and received at least 1 dose of study medication during the long-term extension period
Measure: Number; unit: Participants
Groups:
- Abatacept 30/10 mg/kg: Short-term period: Abatacept 30/10 mg/kg regimen by intravenous (IV) infusion: abatacept 30 mg/kg (by weight) on Days 1, 15, 29, and 57, followed by abatacept (fixed dose) approximating 10 mg/kg on Days 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral Mycophenolate mofetil (MMF) and oral prednisone or prednisone-equivalent Long-term extension period:Participants received abatacept in a weight-tiered dose of approximately 10 mg/kg administered every 28 days by IV infusion in addition to oral MMF and oral prednisone or prednisone-equivalent.
- Abatacept 10/10 mg/kg: Short-term period: Abatacept 10/10 mg/kg regimen by IV infusion: abatacept (fixed dose) approximating 10 mg/kg on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent Long-term extension period:Participants received abatacept in a weight-tiered dose of approximately 10 mg/kg administered every 28 days by IV infusion in addition to oral MMF and oral prednisone or prednisone-equivalent.
- Placebo: Short-term period: Placebo (Dextrose 5% in water [D5W]) or Normal Saline (NS) Short-term period: by IV infusion on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent Long-term extension period:Participants received abatacept in a weight-tiered dose of approximately 10 mg/kg administered every 28 days by IV infusion in addition to oral MMF and oral prednisone or prednisone-equivalent.
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 69 | 66 | 74
Participants
  Day 365 | 43 | 39 | 42
  Day 645 (n=59, 59, and 62) | 45 | 29 | 36

36. Secondary Outcome: Mean Change From Baseline in SLICC/ACR Damage Index
Description: SLICC=Systemic Lupus International Collaborating Clinics; ACR=American College of Rheumatology. The SLICC/ACR Damage Index measures organ damage (nonreversible change, unrelated to active inflammation) occurring since onset of lupus, ascertained by clinical assessment and present for at least 6 months unless otherwise stated. The index assesses 47 items in 12 systems: Ocular, Neuropsychiatric, Renal, Pulmonary, Cardiovascular, Gastrointestinal, Peripheral Vascular, Musculoskeletal, Skin, Premature Gonadal Failure, Diabetes, Malignancy. Scores range from 0 to 2, and the same lesion cannot be scored twice. If damage is noted for a particular item, it is scored 1. No damage is scored 0. Some items may score 2 points if they occur more than once, so that the maximum possible score is 47. Scores can only increase with time, but scores rarely reach over 12. It is usually completed (or updated) yearly.
Time Frame: Day 365 to termination of the long-term extension phase
Population: All randomized participants who received treatment. Treated participants with both post-baseline and baseline measurements showing non-reversible changes in the SLICC/ACR Damage Index (i.e, Change from baseline greater than or equal to 0). 99, 99 and 100 participants were treated respectively. Refer to outcome measure 11 for baseline values
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Abatacept 30/10 mg/kg: Short-term period: Abatacept 30/10 mg/kg regimen by IV infusion: abatacept 30 mg/kg (by weight) on Days 1, 15, 29, and 57, followed by abatacept approximating 10 mg/kg on Days 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent Long-term extension period: Participants received abatacept in a weight-tiered dose of approximately 10 mg/kg administered every 28 days by intravenous (IV) infusion in addition to oral mycophenolate mofetil (MMF) and oral prednisone or prednisone-equivalent.
- Abatacept 10/10 mg/kg: Short-term period: Abatacept 10/10 mg/kg regimen by IV infusion: abatacept approximating 10 mg/kg on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent Long-term extension period: Participants received abatacept in a weight-tiered dose of approximately 10 mg/kg administered every 28 days by intravenous (IV) infusion in addition to oral mycophenolate mofetil (MMF) and oral prednisone or prednisone-equivalent.
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 70 | 67 | 74
Units on a scale
  Day 365 (n=69, 65, 74) | -0.12 (0.06) | -0.17 (0.09) | -0.08 (0.07)
  Day 729 (n=66, 65, 69) | -0.21 (0.10) | -0.28 (0.09) | -0.10 (0.08)
  Day 1093 (n=41, 38, 44) | -.27 (0.13) | -0.16 (0.10) | 0.02 (0.08)

37. Secondary Outcome: Number of Participants With Death, Serious Adverse Events (SAE), Treatment-related Adverse Events SAEs, Discontinuations Due to SAEs, Adverse Events (AEs), Treatment-related AEs, and Discontinuations Due to AEs During Long-term Extension Period
Description: as for outcome 21
Time Frame: From start of study drug in long-term period (Day 365) to up to 56 days after the last dose of the long-term extension (LTE). Deaths in LTE reported to >56 days post last dose.
Population: All participants who entered and received at least 1 dose of study medication during the long-term extension period
Measure: Number; unit: Participants
Groups:
- Abatacept 10 mg/kg: Participants received abatacept in a weight-tiered dose of approximately 10 mg/kg administered every 28 days by intravenous (IV) infusion in addition to oral mycophenolate mofetil (MMF) and oral prednisone or prednisone-equivalent.
Arm/Group | Abatacept 10 mg/kg
Number analyzed (Participants) | 211
Participants
  Deaths | 5
  SAEs | 32
  Treatment-related SAEs | 14
  Discontinuations due to SAEs | 5
  AEs | 183
  Treatment-related AEs | 100
  Discontinuations due to AEs | 10

38. Secondary Outcome: Number of Participants With a Treatment-emergent Seropositive Result During the Long-term Extension Period
Description: Collected in at least 1 sample. Assessment includes immunogenicity (detection of serum antibodies which bind to CTLA4-Ig in the in vitro assays) and exposure to corticosteroids
Time Frame: Day 365 to end of long-term extension period
Population: Immunogenicity analysis population consisted of participants who received at least 1 dose of abatacept and had at least 1 immunogenicity result available.
Measure: Number; unit: Participants
Arm/Group | Abatacept 10 mg/kg
Number analyzed (Participants) | 209
Participants | 17

39. Secondary Outcome: Number of Participants Achieving Renal Response
Description: Renal response=serum creatinine level ≤25% above baseline value and greater than or equal to 50% improvement in the urine protein/creatinine ratio with 1 of the following: urine protein/creatinine ratio (UPCR) <113 mg/mmol, if the baseline ratio was <= 339 mg/mmol OR UPCR <339 mg/mmol,if the baseline ratio >339 mg/mmol.
Time Frame: At Day 365 (end of short-term period) and Day 645
Population: All randomized participants who received treatment.
Measure: Number; unit: participants
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Number analyzed (Participants) | 9 | 66 | 74
participants
  Day 365 | 46 | 66 | 74
  Day 645 (n=59, 59, 62) | 47 | 59 | 62

40. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities During the Long-term Extension Period
Description: preRX=pretreatment; LLN=lower limit of normal; ULN=upper limit of normal. Hemoglobin (g/dL): >3g/dL decrease from preRX value. Hematocrit(%): <0.75*preRX. Erythrocytes (*10^6 c/uL): <0.75*preRX. Platelet count (*10^9 c/L): <0.67*LLN, or >1.5*ULN, or if preRX <LLN, use <0.5*preRX and <100,000/mm^3. Leukocytes (*10^3 c/uL): <0.75*LLN or >1.25*ULN, or if preRX <LLN, use <0.8* preRX or >ULN; if preRX>ULN, use >1.2*preRX or <LLN. Neutrophils + Bands (absolute) (*10^3 c/uL): If value <1.0*10^3 or if value >7.50*10^3 c/uL. Monocytes (absolute) (*10^3 c/uL): If value >2000/mm^3. Basophils (absolute)(*10^3 c/uL): If value >.750*10^3 c/uL. Eosinophils (absolute) (*10^3 c/uL): If value >.750*10^3 c/uL. ALP (U/L): >2*ULN, or if preRX>ULN, use >3* preRX. AST (U/L): >3*ULN, or if preRX>ULN, use >4*preRX. ALT (U/L): >3*ULN, or if preRX>ULN, use >4*preRX. GGT (U/L):>2*ULN, or if preRX >ULN, use >3*preRX. Bilirubin, total (mg/dL): >2*ULN, or if preRX>ULN, use >4*preRX. BUN (mg/dL): >1.5*preRX.
Time Frame: From start of study drug on Day 365 up to 56 days after last dose in the long-term extension period
Population: All participants who entered and received at least 1 dose of study medication during the long-term extension period
Measure: Number; unit: Participants
Arm/Group | Abatacept 10 mg/kg
Number analyzed (Participants) | 211
Participants
  Hemoglobin (low) | 13
  Hemoglobin (high) | NA — Not evaluated
  Hematocrit (n=210) (low) | 11
  Hematocrit (n=210) (high) | NA — Not evaluated
  Erythrocytes (low) | 10
  Erythrocytes (high) | NA — Not evaluated
  Platelet count (n=210) (low) | 1
  Platelet count (n=210) (high) | 0
  Leukocytes (low) | 40
  Leukocytes (high) | 9
  Neutrophils + Bands (absolute) (low) | 4
  Neutrophils + Bands (absolute) (high) | NA — Not evaluated
  Lymphocytes (absolute) (low) | 59
  Lymphocytes (absolute) (high) | 0
  Monocytes (absolute) (low) | NA — Not evaluated
  Monocytes (absolute) (high) | 0
  Basophils (absolute) (low) | NA — Not evaluated
  Basophils (absolute) (high) | 0
  Eosinophils (absolute) (low) | NA — Not evaluated
  Eosinophils (absolute) (high) | 8
  Alkaline phosphatase (ALP) (low) | NA — Not evaluated
  ALP (high) | 3
  Aspartate aminotransferase (AST) (low) | NA — Not evaluated
  AST (high) | 3
  Alanine aminotransferase (ALT) (low) | NA — Not evaluated
  ALT (high) | 5
  G-glutamyl transferase (GGT) (low) | NA — Not evaluated
  GGT (high) | 14
  Bilirubin, total (low) | NA — Not evaluated
  Bilirubin, total (high) | 0
  Blood urea nitrogen (BUN) (low) | NA — Not evaluated
  BUN (high) | 9
  Creatinine (low) | NA — Not evaluated
  Creatinine (high) | 16

41. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities During the Long-term Extension Period (Continued)
Description: LLN=lower limit of normal; ULN=upper limit of normal; preRX=pretreatment. Sodium, serum (mEq/L): <0.95*LLN or >1.05*ULN, or if preRX<LLN, use <0.95*preRX or >ULN if preRX>ULN, use >1.05*preRX or <LLN. Potassium, serum (mEq/L): <0.9* LLN or >1.1*ULN, or if preRX <LLN, use <0.9*preRX or >ULN if preRX>ULN, use >1.1*preRX or <LLN. Chloride, serum (mEq/L): <0.9*LLN or >1.1*ULN, or if preRX<LLN, use <0.9*preRX or >ULN. Calcium, total (mg/dL): <0.8*LLN or >1.2*ULN, or if preRX<LLN, use <0.75*preRX or >ULN if preRX>ULN, use >1.25*preRX or <LLN. Glucose, serum (mg/dL): <65 mg/dL, or >220 mg/dL. Glucose, fasting serum (mg/dL): <0.8*LLN or >1.5*ULN, or if preRX <LLN, use <0.8*preRX or >ULN if preRX>ULN, use >2.0*preRX or <LLN. Albumin (g/dL): <0.9*LLN, or if preRX <LLN, use <0.75*preRX. Cholesterol, total (mg/dL): >2*preRX. Triglycerides (mg/dL): >=2.5*ULN, or if preRX>ULN, use >=2.5*preRX. Triglycerides, fasting (mg/dL): >=2*ULN, or if preRX>ULN, use >2.0*preRX.
Time Frame: From start of study drug on Day 365 up to 56 days after last dose in the long-term extension period
Population: All participants who entered and received at least 1 dose of study medication during the long-term extension period
Measure: Number; unit: Participants
Arm/Group | Abatacept 10 mg/kg
Number analyzed (Participants) | 211
Participants
  Sodium, serum (low) | 1
  Sodium, serum (high) | 2
  Potassium, serum (n=210) (low) | 11
  Potassium, serum (n=210) (high) | 3
  Chloride, serum (low) | 0
  Chloride, serum (high) | 0
  Calcium, total (n=210) (low) | 1
  Calcium, total (n=210) (high) | 2
  Glucose, serum (low) | 23
  Glucose, serum (high) | 2
  Glucose, fasting serum (low) (n=143) | 2
  Glucose, fasting serum (high) (n=143) | 2
  Protein, total (low) | 19
  Protein, total (high) | 0
  Albumin (low) | 12
  Albumin (high) | NA — Not evaluated
  Cholesterol, total (low) (n=32) | 32
  Cholesterol, total (high) (n=32) | NA — Not evaluated
  Triglycerides (low) (n=20) | 20
  Triglycerides (high) (n=20) | NA — Not evaluated
  Triglycerides, fasting (low) (n=18) | 18
  Triglycerides, fasting (high) (n=18) | NA — Not evaluated
  Protein, urine (low) | NA — Not evaluated
  Protein, urine (high) | 9
  Glucose, urine (low) | NA — Not evaluated
  Glucose, urine (high) | 1
  Blood, urine (low) | NA — Not evaluated
  Blood, urine (high) | 35
  Leukocyte esterase, urine (low) (n=185) | NA — Not evaluated
  Leukocyte esterase, urine (high) (n=185) | 27

42. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities During the Long-term Extension Period (Continued)
Description: preRX=pretreatment. Protein, urine: If missing preRX, use >=2, or if value >=4, or if preRX =0 or 0.5, use >=2, or if preRX=1, use >=3, or if preRX=2 OR 3 then use >=4. Glucose, urine: If missing preRX, use >=2, or if value >=4, or if preRX=0 or 0.5, use >=2, or if preRX=1, use >=3, or if preRX=2 or 3, use >=4. Blood, urine: If missing preRX, use >=2, or if value >=4, or if preRX =0 or 0.5, use >=2, or if preRX=1, use >=3, or if preRX=2 or 3, use >=4. Leukocyte esterase, urine: If missing preRX, use >=2, or if value >=4, or if preRX=0 or 0.5, use >=2, or if preRX=1, use >=3, or if preRX=2 or 3, use >=4.
Time Frame: From start of study drug on Day 365 to up to 56 days after last dose in the long-term extension period
Population: All participants who entered and received at least 1 dose of study medication during the long-term extension period
Measure: Number; unit: Participants
Arm/Group | Abatacept 10 mg/kg
Number analyzed (Participants) | 211
Participants
  Protein, urine (low) | NA — Not evaluable
  Protein, urine (high) | 9
  Glucose, urine (low) | NA — Not evaluable
  Glucose, urine (high) | 1
  Blood, urine (low) | NA — Not evaluable
  Blood, urine (high) | 35
  Leukocyte esterase, urine (low) (n=185) | NA — Not evaluable
  Leukocyte esterase, urine (high) (n=185) | 27

ADVERSE EVENTS:
Time Frame: Day 1 of Double-blind Period to within 56 days after last infusion of Double-blind Period or first infusion of Open-label Period, whichever occurred first.
Groups:
- Abatacept 30/10 mg/kg: Abatacept 30/10 mg/kg regimen by intravenous (IV) infusion: In the double-blind period, participants received abatacept 30 mg/kg (by weight) on Days 1, 15, 29, and 57. In the open-label period, participants received abatacept (fixed dose) approximating 10 mg/kg on Days 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral Mycophenolate mofetil (MMF) and oral prednisone or prednisone-equivalent
- Abatacept 10/10 mg/kg: Abatacept 10/10 mg/kg regimen by IV infusion: Participants received abatacept (fixed dose) approximating 10 mg/kg on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 in addition to oral MMF and oral prednisone or prednisone-equivalent.
Arm/Group | Abatacept 30/10 mg/kg | Abatacept 10/10 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 33/99 | 28/99 | 31/100
Other Adverse Events (participants affected / at risk) | 83/99 | 75/99 | 84/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept 30/10 mg/kg (N=99) | Abatacept 10/10 mg/kg (N=99) | Placebo (N=100)
GASTROENTERITIS (Infections and infestations) | 5 | 1 | 2
PNEUMONIA (Infections and infestations) | 4 | 4 | 3
HERPES ZOSTER (Infections and infestations) | 3 | 6 | 0
CELLULITIS (Infections and infestations) | 1 | 1 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 1 | 0
CRYPTOCOCCOSIS (Infections and infestations) | 1 | 0 | 1
JOINT ABSCESS (Infections and infestations) | 1 | 0 | 1
LUNG INFECTION (Infections and infestations) | 1 | 0 | 1
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 | 0 | 0
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 1 | 0 | 0
LOCALISED INFECTION (Infections and infestations) | 1 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
PARONYCHIA (Infections and infestations) | 1 | 0 | 0
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 1 | 0 | 0
PNEUMONIA BACTERIAL (Infections and infestations) | 1 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 1 | 0 | 0
TUBO-OVARIAN ABSCESS (Infections and infestations) | 1 | 0 | 0
UROSEPSIS (Infections and infestations) | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 2 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 2
LUNG ABSCESS (Infections and infestations) | 0 | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 0 | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 1 | 0
TUBERCULOSIS (Infections and infestations) | 0 | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 0 | 2
CANDIDIASIS (Infections and infestations) | 0 | 0 | 1
HISTOPLASMOSIS DISSEMINATED (Infections and infestations) | 0 | 0 | 1
MALARIA (Infections and infestations) | 0 | 0 | 1
MENINGITIS (Infections and infestations) | 0 | 0 | 1
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 1
OTITIS MEDIA CHRONIC (Infections and infestations) | 0 | 0 | 1
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 | 0 | 1
SEPSIS (Infections and infestations) | 0 | 0 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 2 | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 1 | 2
LUPUS NEPHRITIS (Renal and urinary disorders) | 1 | 1 | 0
NEPHRITIS (Renal and urinary disorders) | 1 | 0 | 2
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 0 | 0
GLOMERULONEPHRITIS CHRONIC (Renal and urinary disorders) | 0 | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0
GLOMERULONEPHRITIS (Renal and urinary disorders) | 0 | 0 | 1
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 0 | 0 | 1
MYOCARDITIS (Cardiac disorders) | 2 | 0 | 0
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 1
PYREXIA (General disorders) | 1 | 0 | 2
INFUSION RELATED REACTION (General disorders) | 1 | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 1 | 0 | 1
GENERALISED OEDEMA (General disorders) | 1 | 0 | 0
DRUG INEFFECTIVE (General disorders) | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
CHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0
THROMBOTIC MICROANGIOPATHY (Blood and lymphatic system disorders) | 1 | 0 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 1
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1
HAEMOLYTIC URAEMIC SYNDROME (Blood and lymphatic system disorders) | 0 | 0 | 1
PRESYNCOPE (Nervous system disorders) | 1 | 0 | 0
CONVULSION (Nervous system disorders) | 0 | 2 | 0
HEADACHE (Nervous system disorders) | 0 | 1 | 0
EPILEPSY (Nervous system disorders) | 0 | 0 | 1
VASCULITIS GASTROINTESTINAL (Gastrointestinal disorders) | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1
ASCITES (Gastrointestinal disorders) | 0 | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 0 | 1
SCROTAL OEDEMA (Reproductive system and breast disorders) | 1 | 0 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 1 | 0 | 0
DIPLOPIA (Eye disorders) | 1 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
KAPOSI'S SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
HAEMANGIOMA OF LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
HISTIOCYTOSIS HAEMATOPHAGIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
HAEMATOCRIT DECREASED (Investigations) | 0 | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1 | 0
GALLBLADDER POLYP (Hepatobiliary disorders) | 0 | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept 30/10 mg/kg (N=99) | Abatacept 10/10 mg/kg (N=99) | Placebo (N=99)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 30 | 29 | 32
GASTROENTERITIS (Infections and infestations) | 9 | 7 | 3
URINARY TRACT INFECTION (Infections and infestations) | 9 | 10 | 17
BRONCHITIS (Infections and infestations) | 7 | 8 | 11
NASOPHARYNGITIS (Infections and infestations) | 6 | 11 | 7
ORAL CANDIDIASIS (Infections and infestations) | 6 | 2 | 7
HERPES ZOSTER (Infections and infestations) | 5 | 6 | 2
ORAL HERPES (Infections and infestations) | 2 | 6 | 2
PYREXIA (General disorders) | 13 | 6 | 5
OEDEMA PERIPHERAL (General disorders) | 12 | 9 | 16
CHEST PAIN (General disorders) | 6 | 3 | 3
ASTHENIA (General disorders) | 5 | 2 | 4
FATIGUE (General disorders) | 5 | 4 | 4
DIARRHOEA (Gastrointestinal disorders) | 13 | 11 | 19
NAUSEA (Gastrointestinal disorders) | 10 | 8 | 7
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 5 | 6
VOMITING (Gastrointestinal disorders) | 5 | 5 | 8
MOUTH ULCERATION (Gastrointestinal disorders) | 4 | 2 | 5
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 6 | 4
DYSPEPSIA (Gastrointestinal disorders) | 3 | 5 | 2
GASTRITIS (Gastrointestinal disorders) | 3 | 3 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12 | 7 | 8
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 9 | 7 | 17
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 | 1 | 3
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 | 5 | 8
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 2 | 6
HEADACHE (Nervous system disorders) | 21 | 11 | 15
DIZZINESS (Nervous system disorders) | 7 | 5 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 15
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 3
ACNE (Skin and subcutaneous tissue disorders) | 8 | 7 | 4
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 | 4 | 7
ANAEMIA (Blood and lymphatic system disorders) | 6 | 8 | 9
LEUKOPENIA (Blood and lymphatic system disorders) | 6 | 1 | 5
HYPERTENSION (Vascular disorders) | 9 | 9 | 7
INSOMNIA (Psychiatric disorders) | 5 | 6 | 9
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 4 | 6
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1 | 4 | 6
CONJUNCTIVITIS (Eye disorders) | 0 | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication